CLINICAL TRIAL: NCT03672799
Title: Efficacy of the Rehabilitation Planning Consult for Survivors of Head and Neck Cancer: A Phase II Randomized Controlled Trial
Brief Title: Rehabilitation Planning Consult Phase II Trial
Acronym: RPC-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-5930
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and neck cancer; Rehabilitation; Rehabilitation planning consult; Self-management
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two arms, the experimental arm (Rehabilitation Planning Consult; RPC) and a wait list control (WLC) arm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessor, study investigators, and statistician will remain blinded to group allocation.
  Participants and the treating therapist (Rehabilitation Consultant) will remain unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Planning Consult (RPC) (Experimental): The RPC is a trans-disciplinary, consultative intervention. In the RPC, individualized rehabilitation needs are established, goals are set, strategies to achieve the goals are developed, and follow-through with strategies and goal attainment is facilitated by a rehabilitation professional who consults and collaborates with the survivor. The Rehabilitation Consultant does not provide hands-on treatment, but rather determines the survivors' priority individualized rehabilitation goals, and then helps devise a plan for the survivor to meet those goals independently.
  Participants allocated to RPC will receive a 1 hour consultation with the Rehabilitation Consultant and second consultation 2 to 12 weeks later.
  Interventions: Behavioral: Rehabilitation Planning Consult (RPC)
- Wait list control (WLC) (Active Comparator): There is no standard rehabilitation care for survivors of head and neck cancer at the Princess Margaret Cancer Centre.
  Participants allocated to WLC will enter a 12 week waiting period after which they will crossover to the RPC group.
  Interventions: Behavioral: Rehabilitation Planning Consult (RPC); Other: Wait list control (WLC)

INTERVENTIONS:
Behavioral: Rehabilitation Planning Consult (RPC) — Participants allocated to RPC will receive a 1 hour consultation with the Rehabilitation Consult and second consultation over the next 12 weeks as needed.
  Participants will be assessed at three time points, 1) Baseline assessment, 1 week prior to RPC, 2) post-intervention assessment, 1 week after RPC, and 3) follow-up assessment, 13 weeks after RPC.
  Other Names: RPC
Other: Wait list control (WLC) — Participants who are allocated to WLC will complete a 12 week waiting period. At the end of the waiting period, participants will crossover to the RPC group.
  Participants will be assessed at four time points, 1) Baseline assessment, 1 week prior to waiting period, 2) post-waiting period assessment, 1 week after waiting period, 3) post-intervention assessment, 1 week after RPC, and 4) follow-up assessment,13 weeks after RPC.
  Other Names: WLC
  Arms: Wait list control (WLC)

SUMMARY:
The study will evaluate the efficacy of the Rehabilitation Planning Consult (RPC) to achieve key rehabilitation outcomes in survivors of head and neck cancer compared to a waiting list control group. The RPC is a consultative intervention that teaches survivors to use self-management and problem solving strategies to meet and attain individualized goals. Follow-through with plans and goal attainment are facilitated by a Rehabilitation Consultant. Results from this study will be used to plan for a larger multi-site trial and subsequent real world implementation.

DETAILED DESCRIPTION:
Survivors of head and neck cancer (HNC) often have significant impairments, functional limitations, and reduced quality of life (QL). Rehabilitation services, such as speech-language pathology to improve swallowing, physiotherapy to improve neck mobility, and occupational therapy to enable return to work, can effectively reduce the impact of impairments, restore function, and improve QL. However, access to rehabilitation for survivors of HNC is extremely limited. A trans-professional self-management program is needed to provide resources, links to community providers, and instruction in problem-solving strategies. The program should fit seamlessly into the cancer care system with minimal additional resources. To meet these specifications, an innovative intervention, the Rehabilitation Planning Consult (RPC), was developed and evaluated. The RPC is delivered in 1 to 2 sessions and, in a single arm pilot study, had a moderate to large effect on several aspects of QL and individualized goal attainment. It remains unknown whether the RPC is efficacious in comparison to standard care. In preparation for a Phase III trial, the effect of the RPC, as compared to a standard care control will be estimated, on HNC survivors' QL, attainment of individualized goals, and self-efficacy related to self-management. To facilitate recruitment and ensure ethical provision of services, participants will be randomized to a waiting list control (WLC) or RPC. Assessments will be conducted at three time points for the RPC group and four times for the WLC group. Based on pilot data, approximately 43% of the RPC group are expected to achieve a minimal important difference (MID) in QL, thus 56 participants per arm, 112 participants total, will be recruited. The primary outcome will be QL related to physical health, measured using the SF-36 Physical Component Summary Score (PCS). Secondary measures will include individualized goal performance measured using the Brief Rehabilitation Assessment for Survivors of HNC, disease-specific QL measured with the FACT-HN, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of head and neck cancer
* Completed treatment in the past 6 months

Exclusion Criteria:

* Cognitive issues
* Communication issues
* Presence of major comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Change in the 36-Item Short Form Health Survey - Physical Composite Summary | RPC: 1) 1 week pre-intervention; 2) 1 week post intervention; WLC: 1) 1 week pre-waiting period; 2) 1 week post-waiting period.
  The 36-Item Short Form Health Survey (SF-36) is a self-report generic quality of life measure. The SF-36 has eight domains with scores ranging from 0 to 100, higher scores indicate greater self-reported quality of life. The proportion of participants achieving minimal important difference on the Physical Composite Summary score in the RPC group and WLC group will be analyzed.

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy - Head and Neck scores | RPC: 1) 1 week pre-intervention; 2) 1 week post intervention; WLC: 1) 1 week pre-waiting period; 2) 1 week post-waiting period.
  The Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) is a self-report disease-specific quality of life measure. The FACT-H&N covers 5 domains of quality of life: a) physical well being (score range 0-28), b) social/family well being (score range 0-28), c) emotional well being (score range 0-24), d) functional well being (score range 0-28), and e) head and neck cancer subscale (score range 0-40). A total score can be calculated by adding the 5 subscale scores (total score range 0-148). Higher scores indicate greater better outcomes.
Change in Brief Rehabilitation Assessment for Survivors of Head and Neck Cancer scores | RPC: 1) 1 week pre-intervention; 2) 1 week post intervention; WLC: 1) 1 week pre-waiting period; 2) 1 week post-waiting period.
  The Brief Rehabilitation Assessment for Survivors of Head and Neck Cancer (BRASH) is a self-report measure of individualized goal performance. the measure has three domains, performance, satisfaction, and self-efficacy. Scores for each of the three domains range from 0 to 100, higher scores indicate better outcomes.
Change in 36-Item Short Form Health Survey - Mental Composite Summary scores | RPC: 1) 1 week pre-intervention; 2) 1 week post intervention; WLC: 1) 1 week pre-waiting period; 2) 1 week post-waiting period.
  The 36-Item Short Form Health Survey (SF-36) is a self-report generic quality of life measure. The SF-36 has eight domains with scores ranging from 0 to 100, higher scores indicate better outcomes. The Metal Composite Summary score will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jolie Ringash, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided